CLINICAL TRIAL: NCT02055599
Title: Wound Research Database With Clinical Decision Support for Patients With All Wounds
Brief Title: WEMR With Clinical Decision Support for All Wounds
Status: Withdrawn | Type: Observational
Why Stopped: PI departure.
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 13308-1
Record Dates: First submitted 2014-01-31; First posted 2014-02-05 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2016-11

CONDITIONS: Chronic Wounds
Keywords: Wound; Wound Healing; Pressure Ulcers; Chronic Wounds; Clinical Decision Support
MeSH Terms: conditions — Wounds and Injuries; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this project to begin using a wound research database with clinical decision support features at Winthrop University Hospital. A research database is an electronic computer system that is used to collect patient information. Clinical decision support is the ability for a computer system to provide medical assistance to the doctor through alerts and recommendations based on the information entered. The investigators believe that use of a wound clinical decision support tool, much like a drug, will improve healing in patients with chronic wounds (wounds that fail to heal over the course of weeks) and ultimately lower the risk of death and illness caused by these wounds. In order to develop a useful clinical decision support tool, investigators first need to develop a large research database to determine the data points important for wound healing. The investigators will be using the data collected in this study for future research and publication. Data will be reviewed to answer questions important to wound healing and for the purpose of developing the clinical decision support alert system.

After providing informed consent, participants will be asked a series of questions related to their past medical history, and relevant wound data will be collected. Study staff will photograph the wound at baseline, and once per week until the wound is completely healed, or for a duration of six months.

Participants will be expected to return to Winthrop University Hospital for wound follow-up on a regular basis, or as determined by the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Diagnosed with a wound (defined as a break in the integument)
* Must be willing and able to provide written informed consent

Exclusion Criteria:

* Patients with Diabetic Foot Ulcers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients at Winthrop University Hospital with any chronic wound (defined as a break in the integument).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
To answer questions relevant to wound healing. | up to 6 months
  * How does wound pathology relate to wound healing?
  * How do different types of bacterial infections affect wound healing?
  * To determine the etiology of morbidity, mortality and cost in chronic wound patients.
  * How does providing the patient with an individualized data summary and photos of their wound affect wound healing?

SECONDARY OUTCOMES:
Develop new parameters for clinical decision support based on wound data collected. | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harold Brem, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- See also: Related Info — http://complexwoundhealing.org